CLINICAL TRIAL: NCT02839993
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Associative Learning in Older Adults
Brief Title: tDCS Effects on Associative Learning in Older Adults of Retirement Age
Acronym: TRAINSTIM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TRAINSTIM2.A
Record Dates: First submitted 2016-04-05; First posted 2016-07-21 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Older Adults
Keywords: tDCS effects; associative learning
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Anodal tDCS + training (Experimental): Combination of intensive training of picture-word associations (Wernicko task) with anodal stimulation
  Interventions: Device: tDCS; Behavioral: training
- Sham tDCS + training (Sham Comparator): Combination of intensive training of picture-word associations (Wernicko task) with sham stimulation
  Interventions: Device: tDCS; Behavioral: training

INTERVENTIONS:
Device: tDCS
Behavioral: training
  Other Names: intensive training of picture-word associations

SUMMARY:
The aim of this study is to investigate whether a tDCS-accompanied training of audio-visual associative memory leads to a performance improvement in healthy older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age: old-retired (≥66 years).
* Right handedness
* unobtrusive neuropsychological screening

Exclusion Criteria:

* Mild cognitive impairment (MCI) or other neurological diseases.
* History of severe alcoholism or use of drugs.
* Severe psychiatric disorders such as depression, psychosis (if not in remission) and severe untreated medical problems.
* Contraindication for MRI (claustrophobia, metallic implants, ferromagnetic metals in the body, disorders of thermoregulation, pregnant women)

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Performance in a verbal associative learning paradigm under anodal tDCS compared to sham tDCS. | Performance is assessed within 1 day immediately after training period (several learning blocks) compared to sham
  Investigation whether anodal tDCS leads to improved performance accuracy in the Wernicko task compared to sham stimulation.

SECONDARY OUTCOMES:
Functional connectivity predictors | assessed during baseline testing
  Connectivity as measured by resting-state fMRI during baseline as predictors for performance and tDCS responsiveness
Structural predictors | assessed during baseline testing
  Microstructure of white matter (Fractional Anisotropy) as measured by diffusion tensor imaging during baseline as predictors for performance and tDCS responsiveness
Genotyping of learning related polymorphisms | assessed during baseline screening
  To assess predictors of positive reaction to brain stimulation, genotyping of several learning related polymorphisms will be performed.
Other cognitive outcomes: Attention performance | Performance is assessed within 1 day before and after tDCS + training compared to sham
  Digit span forward performance assessed before and after stimulation to test for tDCS effects on attention
Other cognitive outcomes: working memory | Performance is assessed within 1 day before and after tDCS + training compared to sham
  Digit span backwards performance assessed before and after stimulation to test for tDCS effects on working memory

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Floel A, Rosser N, Michka O, Knecht S, Breitenstein C. Noninvasive brain stimulation improves language learning. J Cogn Neurosci. 2008 Aug;20(8):1415-22. doi: 10.1162/jocn.2008.20098. PMID 18303984
- [Background] Breitenstein C, Knecht S. Development and validation of a language learning model for behavioral and functional-imaging studies. J Neurosci Methods. 2002 Mar 15;114(2):173-9. doi: 10.1016/s0165-0270(01)00525-8. PMID 11856568
- [Background] Breitenstein C, Jansen A, Deppe M, Foerster AF, Sommer J, Wolbers T, Knecht S. Hippocampus activity differentiates good from poor learners of a novel lexicon. Neuroimage. 2005 Apr 15;25(3):958-68. doi: 10.1016/j.neuroimage.2004.12.019. PMID 15808996